CLINICAL TRIAL: NCT06470789
Title: Intervention of Shoulder Blood Flow Restriction Training on Shoulder Joint Pain and Function of Judo Athletes
Acronym: whsu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yang Liu (Other)
Responsible Party: Sponsor-Investigator, Yang Liu, doctor, Wuhan Sports University
Organization: Wuhan Sports University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shoulder rehabilitation
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Shoulder Dislocation; Blood Flow Restriction Training
MeSH Terms: conditions — Shoulder Dislocation | interventions — Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- blood flow restriction training (Experimental): blood flow restriction training (BFRT) is a popular method of sports training. It involves the use of devices such as air sleeves or elastic bands with adjustable functions during sports training that restrict blood flow to parts of the limb, resulting in an adaptive effect similar to high-intensity training in the muscles, while actually using relatively light weights. BFRT is usually combined with light exercise, such as low-load strength training or aerobic training, to build muscle strength and muscle endurance. This training method is more friendly to patients after sports injuries ， fractures, joint surgery ， etc. It can help to train the injured area with light loads to reduce muscle atrophy and speed up recovery to restore muscle function and strength. BFRT is also commonly used by athletes in different sports to improve muscle strength and endurance while reducing weight load, helping to reduce the risk of overtraining and injury.
  Interventions: Behavioral: Shoulder blood restriction training
- Massage (Placebo Comparator): Massage is a widely used traditional Chinese physical therapy technique, which uses massage, kneading, pushing, flicking, tapping and other techniques, as well as the use of the palm, fingertips, elbows, knees and other body parts to stimulate specific body areas or acupoints to achieve the purpose of treatment or relief of disease symptoms . Massage massage can relieve musculoskeletal pain by promoting blood circulation, relaxing tense muscles and reducing inflammation, and improve muscle elasticity and flexibility, helping to reduce muscle tension and stiffness . Therefore, massage massage is often used to improve the treatment of local body pain, and a large number of studies have shown that massage massage can reduce shoulder pain in the short term, restore shoulder function and improve the range of motion of shoulder joints .
  Interventions: Behavioral: Shoulder blood restriction training
- BFRT combined massage group (Experimental): To observe the effect of blood flow restriction equipment combined with low-load shoulder resistance training and massage intervention on shoulder pain, function, strength and joint motion of judo athletes with shoulder joint dysfunction.
  Interventions: Behavioral: Shoulder blood restriction training

INTERVENTIONS:
Behavioral: Shoulder blood restriction training — Massage massage is also often used to improve the treatment of local body pain, and a large number of studies have shown that massage massage can reduce shoulder pain in the short term, restore shoulder function and improve the range of motion of shoulder joints.
  Other Names: massage

SUMMARY:
To observe the effect of shoulder low load blood flow restriction training on pain, function, strength and joint motion of the subjects with shoulder joint dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* ① Judo athletes, aged 18-30 years old; ② can cooperate with rehabilitation physiotherapy and training and follow-up, and will not quit the study without reason; The presence of shoulder joint pain and dysfunction; After passing the shoulder function test screening, there are two or more positive tests

Exclusion Criteria:

* External injuries of shoulder joint, including bumps, blows, cuts, burns, contusions, etc., without skin rupture, external blood or subcutaneous bleeding; ② congenital abnormal bone structure; ③ There is inflammation, dislocation of shoulder joint, ligament injury; ④ A history of shoulder joint related surgery within one year; ⑤ Injury or discomfort to other body parts;

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Shoulder strength | 6week
  In this study, a muscle force tester was used to measure the maximum force of the subjects' shoulders. During the measurement, the subjects were required to maintain supine and standing positions, and the maximum force of shoulder joint push, abduction, internal rotation and external rotation was measured in different positions. The strength test of each exercise session needs to be completed three times, each measurement interval of 30 seconds, and finally the average value of the three maximum strength values is taken.
Shoulder joint range of motion Angle measurement | 6week
  The measurement of shoulder joint range of motion mainly includes measuring the range Angle of shoulder joint abduction, external rotation and internal rotation under different postures (standing posture, supine posture).
Shoulder VAS score | 6week
  In this study, the quantification of shoulder joint pain was carried out using the Visual Analogue Scale (VAS) . VAS is a common tool used to assess the level of pain or discomfort, including shoulder pain.
Shoulder Constant-Murley scale | 6week
  Shoulder Constant-Murley scale is a clinical evaluation tool used to evaluate shoulder function and severity of shoulder diseases, and is often used to evaluate the efficacy and rehabilitation progress before and after shoulder surgery. The scale includes assessments of shoulder joint range of motion, muscle strength, pain and function of daily living.

CONTACTS AND LOCATIONS:
Locations (1):
- YangLiu, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
It involves personal privacy